CLINICAL TRIAL: NCT04401163
Title: Long-term Pulmonary Outcomes After Infection With Sars-CoV-2
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 33510
Record Dates: First submitted 2020-05-12; First posted 2020-05-26 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2022-11

CONDITIONS: Sars-CoV2; Covid19
MeSH Terms: conditions — COVID-19 | interventions — Blood Specimen Collection; Respiratory Function Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Imaging of the lungs — After hospital admissions with COVID19 patients will come for two clinical visits to complete a number of questionnaires, pulmonary function testing, six-minute walk test, blood sampling and imaging of the lungs.
  Other Names: Blood sampling; Health related quality of life measurements; Pulmonary function tests

SUMMARY:
The objective of this study is to assess the long-term outcomes after hospital admission with Covid-19 with respect to pulmonary function, physical capacity, imaging, quality of life and socioeconomic outcomes.

DETAILED DESCRIPTION:
Patients will be invited to follow-up visits 3 and 12 months after hospitalization with COVID19.

Inclusion will take place during 2020. We expect to enroll 180 non-ICU patients and 36 ICU patients.

ELIGIBILITY:
Inclusion Criteria:

* Infection with Sars-CoV-2

Exclusion Criteria:

* Unable to attend hospital visits due to frailty or severe disease
* Unable to understand and complete questionnaires due to intellectual or language limitations / deficits

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients hospitalized due to infection with Covid-19 and submitted from any of the five hospitals in the Central Denmark Region will be invited to participate.
Sampling Method: Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2020-06-18 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Imaging of the lungs | 3 months after discharge
  Expert evaluation
Imaging of the lungs | 12 months after discharge
  Expert evaluation
Pulmonary function tests | 3 months after discharge
  Liter
Pulmonary function tests | 12 months after discharge
  Liter
Six-minute walk test | Performed 3 months after discharge
  Walking distance (meters) and change in oxygen saturation.
Six-minute walk test | Performed 12 months after discharge
  Walking distance (meters) and change in oxygen saturation.

SECONDARY OUTCOMES:
Short Form-36 (SF-36) questionnaire | 3 months after discharge
  0-100 scale. The lower the score, the more disability.
Short Form-36 (SF-36) questionnaire | 12 months after discharge
  0-100 scale. The lower the score, the more disability.
Fatigue Assessment Score | 3 months after discharge
  10-50 score. The higher the score, the more fatigue
Fatigue Assessment Score | 12 months after discharge
  10-50 score. The higher the score, the more fatigue
Cognitive sore (MOCA) | 3 months after discharge
  0-30. The lower the score, the more cognitive impairment
Cognitive sore (MOCA) | 12 months after discharge
  0-30. The lower the score, the more cognitive impairment
Hospital anxiety and Depression score (HADS) | 3 months after discharge
  0-21. The higher the score, the more risk of anxiety or depression.
Hospital anxiety and Depression score (HADS) | 12 months after discharge
  0-21. The higher the score, the more risk of anxiety or depression.
Comorbidities | 12 months after discharge
  Any pre-COVID-19 comorbidity and treatment with immmunosuppressants will be registered.
Blood sample at routine follow up. | 3 months after discharge
  Change in outcomes between discharge and follow-up visits will be evaluated
Blood sample at routine follow up. | 12 months after discharge
  Change in outcomes between discharge and follow-up visits will be evaluated
Biobanking of blood | 3 months after discharge
  Knowledge regarding COVID19 is drastically evolving. Biobanking makes it possible to investigate blood samples in the future corresponding to ongoing evidence.
Biobanking of blood | 12 months after discharge
  Knowledge regarding COVID19 is drastically evolving. Biobanking makes it possible to investigate blood samples in the future corresponding to ongoing evidence.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Bendstrup, MD, PhD, Principal Investigator — Aarhus University Hospital
Locations (6):
- Denmark (6):
  - Aarhus University Hospital, Aarhus
  - Regional Hospital, Holstebro, Holstebro
  - Regional Hospital, Horsens, Horsens
  - Regional Hospital, Randers, Randers
  - Regional Hospital, Silkeborg, Silkeborg
  - Regional Hospital, Viborg, Viborg

IPD SHARING:
Plan to Share IPD: Undecided